CLINICAL TRIAL: NCT05204745
Title: Gait and Balance Impairment, Dementia and Wide Brain Ventricles in the Ages 65-84 Years
Brief Title: Ventriculomegaly and Gait Disturbance in the Senior Population in the Region of Västerbotten
Acronym: VESPR
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Principal Investigator, Jan Malm, MD, PhD, Umeå University
Other Study IDs: 2017/335-31
Record Dates: First submitted 2021-10-01; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH); Brain Diseases; Central Nervous System Diseases; Dementia; Gait Disorders, Neurologic; Hydrocephalus, Normal Pressure
Keywords: Idiopathic Normal Pressure Hydrocephalus
MeSH Terms: conditions — Brain Diseases; Central Nervous System Diseases; Dementia; Gait Disorders, Neurologic; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Subjects with subjective gait impariment according to questionnaire answers.
- Control: Subjects without subjective gait impariment according to questionnaire answers.

SUMMARY:
Idiopathic normal pressure hydrocephalus (INPH) is a treatable disease of the elderly, typically causing gait impariment, dementia and urinary incontinence. The objective of this study is to make an epidemiological survey of INPH in Umeå, Sweden. Subjects with self-perceived gait impairments will be identified through a questionnaire. They will go through clinical examinations and have an MRI of the brain. A control population will also be investigated to enable comparisons between the populations. The main hypothesis is that the prevalence of INPH in the population is higher than what is previoulsy known.

ELIGIBILITY:
Inclusion Criteria:

- Living in Umeå, Sweden.

Exclusion Criteria:

* Age <65 or >84 years when the questionnaire was sent out.
* Death at the time for the clinical evaluation.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The number of people, aged 65-84 years and living in Umeå, is approximately 18 000. Of these, 6500 will be randomly selected from the Swedish population registry. They will be asked to answer a mailed-out questionnaire regarding self-perceived gait impairment. Those with self-percieved gait impairment will be invited for clinical examinations as cases and a random selection of those without self-percieved gait impairment will be invited to participate in clinical examinations as controls.
Sampling Method: Probability Sample
Enrollment: 6500 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with Idiopathic Normal Pressure Hydrocephalus | Through study completion, an average of approximately 1 month.
  Diagnosis of INPH based on clinical evaluation and MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Norrlands Universitetssjukhus, Umeå, Västerbotten County, Sweden